CLINICAL TRIAL: NCT05579977
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND, PLACEBO CONTROLLED, DOSE RANGING, DOSE FINDING, PARALLEL GROUP STUDY TO ASSESS EFFICACY AND SAFETY OF PF-07081532, AND OPEN LABEL ORAL SEMAGLUTIDE, IN ADULTS WITH TYPE 2 DIABETES MELLITUS (T2DM) INADEQUATELY CONTROLLED ON METFORMIN, AND SEPARATELY PF-07081532 COMPARED TO MATCHING PLACEBO IN ADULTS WITH OBESITY BUT WITHOUT T2DM
Brief Title: Trial to Learn About the Study Medicine (PF-07081532) and Rybelsus in People With Type 2 Diabetes and Separately PF-07081532 in People With Obesity
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The decision to terminate clinical development of PF-07081532 is based on pharmacokinetic data from Phase 1 drug-drug-interaction studies and laboratory measurements of elevated transaminases in these Phase 1 studies as well as a Phase 2 study.
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: C3991004; 2022-002834-15 (EudraCT Number)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Results first posted 2024-08-01 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Diabetes Mellitus; Obesity
Keywords: Diabetes Mellitus; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Obesity | interventions — semaglutide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- PF-07081532 20 mg T2DM (Experimental): PF-07081532 20 mg daily in T2DM
  Interventions: Drug: PF-07081532
- PF-07081532 40 mg T2DM (Experimental): PF-07081532 40 mg daily in T2DM
  Interventions: Drug: PF-07081532
- PF-07081532 80 mg T2DM (Experimental): PF-07081532 80 mg daily in T2DM
  Interventions: Drug: PF-07081532
- PF-07081532 160 mg T2DM (Experimental): PF-07081532 160 mg daily in T2DM
  Interventions: Drug: PF-07081532
- PF-07081532 260 mg T2DM (Experimental): PF-07081532 260 mg daily in T2DM
  Interventions: Drug: PF-07081532
- Placebo T2DM (Placebo Comparator): Placebo daily in T2DM
  Interventions: Other: Placebo
- PF-07081532 80 mg Obesity (Experimental): PF-07081532 80 mg daily in Obesity
  Interventions: Drug: PF-07081532
- PF-07081532 140 mg Obesity (Experimental): PF-07081532 140 mg daily in Obesity
  Interventions: Drug: PF-07081532
- PF-07081532 200 mg Obesity (Option 1) (Experimental): PF-07081532 200 mg daily in Obesity
  Interventions: Drug: PF-07081532
- PF-07081532 200 mg Obesity (Option 2) (Experimental): PF-07081532 200 mg daily in Obesity
  Interventions: Drug: PF-07081532
- PF-07081532 260 mg Obesity (Experimental): PF-07081532 260 mg daily in Obesity
  Interventions: Drug: PF-07081532
- Rybelsus 14 mg T2DM (Active Comparator): Semaglutide 14 mg daily in T2DM
  Interventions: Drug: Rybelsus
- Placebo Obesity (Placebo Comparator): Placebo in Obesity
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: PF-07081532 — Oral glucagon-like peptide-1 receptor agonist
  Arms: PF-07081532 140 mg Obesity; PF-07081532 160 mg T2DM; PF-07081532 20 mg T2DM; PF-07081532 200 mg Obesity (Option 1); PF-07081532 200 mg Obesity (Option 2); PF-07081532 260 mg Obesity; PF-07081532 260 mg T2DM; PF-07081532 40 mg T2DM; PF-07081532 80 mg Obesity; PF-07081532 80 mg T2DM
Other: Placebo — No drug
  Arms: Placebo Obesity; Placebo T2DM
Drug: Rybelsus — Oral Semaglutide
  Arms: Rybelsus 14 mg T2DM

SUMMARY:
The purpose of this study is to find out if PF-07081532 ("the active study drug"), is safe and helps treat people with obesity without diabetes to lose weight, and people with diabetes to keep their blood sugar in good control. Individuals diagnosed with diabetes that are on metformin or individuals with obesity without diabetes will be included in the study.

Those participating in the diabetes part of the study, will receive either active study drug, placebo, or an approved treatment called Rybelsus. Those in the obesity part of the study, will receive either active study drug or placebo. The study will last for about 36 weeks except for the first 25% of the participants that enter in which case the study will last for approximately 48 weeks. during this time there will be visits every 4 weeks with phone calls in between.

ELIGIBILITY:
Inclusion Criteria:

T2DM

* T2DM inadequately controlled with metformin
* BMI ≥23.0 kg/m2 (≥20.0 kg/m2 in Japan)
* HbA1C of 7% to 10% (53-86 mmol/mol)
* FPG ≤270 mg/dL (15 mmol/L)

Obesity

* BMI ≥30.0 kg/m2
* HbA1C ≤6.4% (47 mmol/mol)
* FPG ≤126 mg/dL (7 mmol/L)

Exclusion Criteria:

* Any of the following: Active/current, symptomatic gallbladder disease; History of pancreatitis in the prior 2-months;History of Type 1 Diabetes Mellitus, or secondary forms of diabetes; Any condition affecting drug absorption; Medical history of active liver disease (other than non-alcoholic hepatic steatosis)
* Use of pharmacological agents with approved indication for weight loss
* T2DM:Use of any agent (other than metformin)for the explicit purpose of glycemic control;History of diabetic ketoacidosis;Proliferative retinopathy or maculopathy requiring acute treatment;
* Obesity: Previous or planned weight reduction surgery; Major depressive disorder or other severe psychiatric disorders; Any lifetime history of a suicide attempt; PHQ-9 score ≥15; Response of "yes" to Question 4 or 5, or on any suicidal behavioral question on the C-SSRS
* Clinically significant cardiovascular conditions
* Uncontrolled blood pressure
* Personal or within first-degree relative family history of MTC or MEN2
* Other medical or psychiatric condition that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study
* Any of the following central lab results: Fasting C-peptide <0.8 ng/mL; ALT or AST ≥2.5x ULN; Direct bilirubin >ULN or T Bili >1.5x ULN except when participants have a history of Gilbert syndrome ; TSH >1.5x ULN or <LLN; Serum calcitonin >ULN; Serum amylase or serum lipase >ULN; eGFR <45 ml/min/1.73 ; Active Hepatitis B, or Hepatitis C; A positive urine drug test for illicit drugs

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 902 (Actual)
Dates: Start 2022-10-27 (Actual); Primary Completion 2023-07-14 (Actual); Study Completion 2023-09-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (88):
- United States (39):
  - Trinity Clinical Research, Centreville, Alabama
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - San Fernando Valley Health Institute, Canoga Park, California
  - Catalina Research Institute, LLC, Montclair, California
  - Empire Clinical Research, Pomona, California
  - University Clinical Investigators, Inc., Tustin, California
  - Diablo Clinical Research, Inc., Walnut Creek, California
  - Innovative Research of West Florida, Clearwater, Florida
  - Jacksonville Center for Clinical Research, Jacksonville, Florida
  - Adult Medicine of Lake County, Mt. Dora, Florida
  - Endocrine Research Solutions, Inc., Roswell, Georgia
  - Cedar Crosse Research Center, Chicago, Illinois
  - Evanston Premier Healthcare Research LLC, Skokie, Illinois
  - Iowa Diabetes and Endocrinology Research Center, West Des Moines, Iowa
  - Anderson Medical Research, Ft. Washington, Maryland
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Mercury Street Medical Group, PLLC, Butte, Montana
  - Hassman Research Institute, Berlin, New Jersey
  - Premier Research, Trenton, New Jersey
  - Medication Management, Greensboro, North Carolina
  - Meridian Clinical Research, LLC, Cincinnati, Ohio
  - Alliance for Multispecialty Research, LLC, Norman, Oklahoma
  - Heritage Valley Multispecialty Group, Inc, Beaver, Pennsylvania
  - Preferred Primary Care Physicians, Preferred Clinical Research (Ofc 18), Pittsburgh, Pennsylvania
  - Preferred Primary Care Physicians, Uniontown, Pennsylvania
  - Velocity Clinical Research, Providence, East Greenwich, Rhode Island
  - HealthStar Physicians, P.C., Morristown, Tennessee
  - Healthstar Physicians, Morristown, Tennessee
  - Elligo Clinical Research Center, Austin, Texas
  - Velocity Clinical Research, Dallas, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - Medical Colleagues of Texas, LLP, Katy, Texas
  - Tapia Internal Medicine Clinic, Paris, Texas
  - Northeast Clinical Research of San Antonio, San Antonio, Texas
  - Consano Clinical Research, LLC, Shavano Park, Texas
  - Sugar Lakes Family Practice, Sugar Land, Texas
  - Chrysalis Clinical Research, St. George, Utah
  - Southwest Internal Medicine, St. George, Utah
  - Manassas Clinical Research Center, Manassas, Virginia
- Bulgaria (5):
  - Medical Centre "Asklepiy", Dupnitsa, Kyustendil
  - MHAT Botevgrad, Botevgrad, Sofia
  - Diagnostic Consultative Center Aleksandrovska, Sofia, Sofia (stolitsa)
  - Medical Center Zdrave 1, Kozloduy, Vratsa
  - "Prevencia - 2000 - Medical Center for Prehospital Medical Care" OOD, Stara Zagora
- Canada (11):
  - Dr. M.B. Jones Inc., Victoria, British Columbia
  - G A Research Associates, Moncton, New Brunswick
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Dawson Clinical Research, Guelph, Ontario
  - Milestone Research Inc., London, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - Manna Research Mirabel, Mirabel, Quebec
  - Diex Recherche Victoriavile Inc., Victoriaville, Quebec
  - Diex Recherche Quebec Inc., Québec
  - Centre de Recherche Saint-Louis, Québec
- Czechia (8):
  - MUDr. Alena Vachova, České Budějovice, Jihočeský kraj
  - EDUMED s.r.o., Broumov, Kralovehradecky KRAY
  - Kardiologicka a Angiologicka Ambulance, Ostrava, Ostrava Město
  - Clinical Trials Service s.r.o., Uherské Hradiště, Zlín
  - Agentura Science Pro, Olomouc
  - Private Practice - Dr. Tomáš Brychta, Olomouc
  - EUC Klinika Praha, Prague
  - Clinical Trials Service s.r.o., Uherské Hradiště
- Hungary (6):
  - Belinus Orvosi és Számitástechnikai Bt, Debrecen, Hajdú-Bihar
  - Borbánya Praxis, Nyíregyháza, Borbánya, Szabolcs-Szatmár-Bereg
  - CLINFAN Szolgáltató Kft, Szekszárd, Tolna County
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - ClinDiab Kft., Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Japan (10):
  - Nakakinen clinic, Naka, Ibaraki
  - Yokohama Minoru Clinic, Yokohama, Kanagawa
  - Shiraiwa Medical Clinic, Kashihara, Osaka
  - Medical Corporation Heishinkai OCROM Clinic, Suita-shi, Osaka
  - Seiwa Clinic, Adachi-ku, Tokyo
  - Tokyo-Eki Center-building Clinic, Chuo-ku, Tokyo
  - Medical Corporation Chiseikai Tokyo Center Clinic, Chuo-ku, Tokyo
  - Fukuwa Clinic, Chuo-ku, Tokyo
  - Medical Corporation Heishinkai ToCROM Clinic, Shinjuku-ku, Tokyo
  - Yokohama Minoru Clinic, Yokohama
- Poland (7):
  - Oświęcimskie Centrum Badań Klinicznych, Oświęcim, Lesser Poland Voivodeship
  - KO-MED Centra Kliniczne Pulawy, Puławy, Lublin Voivodeship
  - Zdrowie Osteo-Medic, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Przychodnia Specjalistyczna Andrzej Wittek, Henryk Rudzki, Ruda Śląska, Silesian Voivodeship
  - Gabinet Lekarski Małgorzata Jadwiga Saryusz-Wolska, Lodz
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan
- Puerto Rico (2):
  - Latin Clinical Trial Center, San Juan
  - GCM Medical Group, PSC - Hato Rey Site, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Amin NB, Frederich R, Tsamandouras N, Haggag AZ, Schuster T, Zmuda W, Palmer A, Vasas S, Buckley G, Smith TR, DuBrava SJ, Zhu Q, Johnson M. Evaluation of an oral small-molecule glucagon-like peptide-1 receptor agonist, lotiglipron, for type 2 diabetes and obesity: A dose-ranging, phase 2, randomized, placebo-controlled study. Diabetes Obes Metab. 2025 Jan;27(1):215-227. doi: 10.1111/dom.16005. Epub 2024 Oct 16. PMID 39415344
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C3991004

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study had 2 cohorts: Cohort 1 included participants with type 2 diabetes mellitus (T2DM) on a background therapy of metformin. Cohort 2 included participants with obesity but without T2DM.
Pre-assignment Details: A total of 902 participants were randomized in this study of which 1 participant did not receive treatment. The study was terminated based on pharmacokinetic data from Phase 1 drug-drug-interaction studies and laboratory measurements of elevated transaminases in these Phase 1 studies as well as this Phase 2 study.
Groups:
- Placebo (T2DM): Participants randomized to receive a single dose of PF-07081532-matching placebo once daily (QD) orally.
- PF-07081532 20mg (T2DM): Participants randomized to receive PF-07081532 20 mg QD orally.
- PF-07081532 40mg (T2DM): Participants randomized to receive PF-07081532 20 mg QD orally for 4 weeks, followed by 40 mg QD orally.
- PF-07081532 80mg (T2DM); PF-07081532 80mg (Obesity): Participants randomized to receive PF-07081532 20 mg QD, 40 mg QD and 60 mg QD orally for 4 weeks, followed by PF-07081532 80 mg QD orally.
- PF-07081532 160mg (T2DM): Participants randomized to receive PF-07081532 20 mg QD 40 mg QD, 60 mg QD, 80 mg QD and 120 mg QD orally for 4 weeks, followed by PF-07081532 160 mg QD orally.
- PF-07081532 260mg (T2DM): Participants randomized to receive PF-07081532 20 mg QD, 40 mg QD, 80 mg QD, 140 mg QD and 200 mg QD orally for 4 weeks, followed by PF-07081532 260 mg QD orally.
- Rybelsus 14mg (T2DM): Participants randomized to receive Rybelsus 3 mg QD and 7 mg QD each for 4 weeks followed by 14 mg QD.
- Placebo (Obesity): Participants randomized to receive a single dose of PF-07081532-matching placebo QD orally.
- PF-07081532 140mg (Obesity): Participants randomized to receive PF-07081532 20 mg QD, 40 mg QD and 60 mg QD, 80 mg QD,120 mg QD orally for 4 weeks each followed by PF-07081532 140 mg QD orally.
- PF-07081532 200mg (Obesity,5 Steps): Participants randomized to receive PF-07081532 20 mg QD, 40 mg QD and 60 mg QD, 100 mg QD,160 mg QD orally for 4 weeks each followed by PF-07081532 200 mg QD orally.
- PF-07081532 200mg (Obesity,4 Steps): Participants randomized to receive PF-07081532 20 mg QD, 40 mg QD and 80 mg QD, 140 mg QD orally for 4 weeks each followed by PF-07081532 200 mg QD orally.
- PF-07081532 260mg (Obesity): Participants randomized to receive PF-07081532 20 mg QD, 40 mg QD and 80 mg QD, 140 mg QD, 200 mg QD orally for 4 weeks each followed by PF-07081532 260 mg QD orally.
Period: Treatment Phase
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM) | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Started | 75 | 73 | 72 | 73 | 73 | 74 | 73 | 64 | 66 | 64 | 65 | 66 | 64
Received Treatment | 75 | 73 | 72 | 73 | 72 | 74 | 73 | 64 | 66 | 64 | 65 | 66 | 64
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 75 | 73 | 72 | 73 | 73 | 74 | 73 | 64 | 66 | 64 | 65 | 66 | 64
Not completed — Other | 0 | 0 | 0 | 2 | 1 | 2 | 1 | 2 | 2 | 1 | 0 | 0 | 3
Not completed — Treatment with restricted medication needed | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 1 | 2 | 0 | 1 | 8 | 3 | 3 | 5 | 1 | 3
Not completed — Study terminated by sponsor | 70 | 70 | 61 | 59 | 63 | 53 | 66 | 48 | 47 | 37 | 44 | 36 | 32
Not completed — Pregnancy | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 1 | 2 | 2 | 1 | 4 | 3
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 11 | 10 | 5 | 17 | 5 | 5 | 12 | 20 | 15 | 24 | 23
Not completed — Randomized not treated | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Period: Follow up
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM) | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Started | 75 (Eligible participants who withdrew from treatment could enter the follow-up phase. 1 participant with withdrawal reason as Death in treatment phase was also counted in follow-up as exact date of last dose was unknown.) | 73 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 72 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 73 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 72 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 74 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 73 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 64 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 66 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 64 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 65 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 66 (Eligible participants who withdrew from treatment could enter the follow-up phase.) | 64 (Eligible participants who withdrew from treatment could enter the follow-up phase.)
Completed | 72 | 73 | 72 | 72 | 70 | 72 | 71 | 59 | 61 | 59 | 60 | 61 | 57
Not Completed | 3 | 0 | 0 | 1 | 2 | 2 | 2 | 5 | 5 | 5 | 5 | 5 | 7
Not completed — Death | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 3 | 2 | 2 | 4 | 4
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 1 | 0 | 1 | 4 | 2 | 3 | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Groups:
- Placebo (T2DM); Placebo (Obesity): Participants randomized to receive a single dose of PF-07081532-matching placebo QD orally.
- Total: Total of all reporting groups
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM) | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity) | Total
Number analyzed (Participants) | 75 | 73 | 72 | 73 | 72 | 74 | 73 | 64 | 66 | 64 | 65 | 66 | 64 | 901
Age, Customized [Count of Participants; unit: Participants]
  Less than (<) 18 years | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  18-44 years | 6 | 8 | 3 | 4 | 4 | 6 | 5 | 17 | 25 | 24 | 25 | 21 | 23 | 171
  45-64 years | 40 | 39 | 52 | 48 | 44 | 36 | 43 | 36 | 33 | 35 | 34 | 39 | 33 | 512
  More than equal to (>=) 65 years | 29 | 26 | 17 | 21 | 24 | 32 | 25 | 11 | 8 | 5 | 6 | 6 | 8 | 218
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 30 | 29 | 31 | 33 | 31 | 36 | 36 | 38 | 45 | 36 | 42 | 40 | 469
  Male | 33 | 43 | 43 | 42 | 39 | 43 | 37 | 28 | 28 | 19 | 29 | 24 | 24 | 432
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 14 | 13 | 8 | 7 | 14 | 10 | 8 | 5 | 8 | 10 | 14 | 12 | 10 | 133
  Not Hispanic or Latino | 61 | 60 | 63 | 66 | 58 | 64 | 64 | 59 | 58 | 54 | 51 | 54 | 54 | 766
  Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 1 | 5
  Asian | 12 | 14 | 17 | 15 | 13 | 14 | 11 | 4 | 3 | 3 | 3 | 4 | 6 | 119
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
  Black or African American | 4 | 2 | 4 | 4 | 5 | 5 | 5 | 4 | 6 | 15 | 6 | 5 | 4 | 69
  White | 58 | 57 | 51 | 54 | 54 | 54 | 57 | 55 | 56 | 44 | 56 | 55 | 52 | 703
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Placebo-adjusted, Change From Baseline in Percentage of Glycated Hemoglobin (HbA1c) at Week 32: Cohort 1 (Type 2 Diabetes Mellitus)
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Placebo-adjusted, Percent Change From Baseline in Body Weight at Week 32: Cohort 2 (Obesity)
Description: Body weight was measured using a calibrated weighing scale.
Time Frame: Baseline (result closest prior to dosing on Day 1), week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Percentage of Participants Who Achieved HbA1C <7% at Week 32: Cohort 1 (Type 2 Diabetes Mellitus)
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 32: Cohort 1 (Type 2 Diabetes Mellitus)
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

5. Secondary Outcome: Percent Change From Baseline in Body Weight at Week 32: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Body weight was measured using a calibrated weighing scale.
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Placebo-adjusted, Change From Baseline in HbA1C in the Rybelsus Arm at Week 32: Cohort 1 (Type 2 Diabetes Mellitus)
Description: This outcome measure was planned to be analyzed only for rybelsus arm and placebo arm as pre-specified in the protocol.
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Percentage of Participants Achieving >=5%, >=10%, and >=15% Body Weight Loss at Week 32 Relative to Baseline: Cohort 2 (Obesity)
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

8. Secondary Outcome: Absolute Change From Baseline in Waist Circumference at Week 32: Cohort 2 (Obesity)
Description: Waist circumference was measured at midpoint, between lower margin of last palpable rib and top of iliac crest (approximately 1 inch [2.54 centimeter {cm}] above the navel). It was measured by using an anthropometric tape (stretch-resistant).
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Absolute Change From Baseline in Waist-to-hip Ratio at Week 32: Cohort 2 (Obesity)
Description: The hip circumference was defined as the circumference around the widest portion of the buttocks. Waist circumference was measured at midpoint, between lower margin of last palpable rib and top of iliac crest (approximately 1 inch [2.54 cm] above the navel). The measurements were performed using an anthropometric tape (stretch-resistant).
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

10. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) at Week 32: Cohort 2 (Obesity)
Description: HOMA-IR was calculated as: fasting plasma insulin ([FPI]*(FPG)/405 and measured in terms of mg/dL* (milliunits per liter).
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

11. Secondary Outcome: Change From Baseline in Homeostatic Model Assessment for Insulin Sensitivity (HOMA-S) at Week 32: Cohort 2 (Obesity)
Description: HOMA-S was calculated as (22.5/[FPI] * FPG) *100 and measured in terms of percentage sensitivity.
Time Frame: Baseline (result closest prior to dosing on Day 1), Week 32
Population: Data was not collected for this outcome measure as the study was terminated prior to any participant reaching Week 32.
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Cohort 1 (Type 2 Diabetes Mellitus)
Description: An adverse event (AE) was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred on or after the first dose of treatment but before the last dose plus lag time.
Time Frame: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 75 | 73 | 72 | 73 | 72 | 74 | 73
Participants | 35 | 37 | 50 | 44 | 45 | 56 | 36

13. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (TEAEs): Cohort 2 (Obesity)
Description: An AE was any untoward medical occurrence in a participant or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. TEAEs were any AEs that occurred on or after the first dose of treatment but before the last dose plus lag time.
Time Frame: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 66 | 64 | 65 | 66 | 64
Participants | 44 | 54 | 50 | 56 | 60 | 53

14. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs): Cohort 1 (Type 2 Diabetes Mellitus)
Description: SAE defined as any untoward medical occurrence that, at any dose, met one or more of the following criteria: resulted in death; was life-threatening; required inpatient hospitalization or prolongation of hospitalization; resulted in persistent or significant disability/incapacity (substantial disruption of the ability to conduct normal life functions); resulted in congenital anomaly/birth defect; was a suspected transmission via a Pfizer product of an infectious agent, pathogenic or non-pathogenic; other important medical events.
Time Frame: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 75 | 73 | 72 | 73 | 72 | 74 | 73
Participants | 1 | 0 | 3 | 3 | 1 | 2 | 1

15. Secondary Outcome: Number of Participants With Serious Adverse Events (SAEs): Cohort 2 (Obesity)
Description: as for outcome 14
Time Frame: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 66 | 64 | 65 | 66 | 64
Participants | 1 | 2 | 2 | 1 | 2 | 2

16. Secondary Outcome: Number of Participants Reporting Adverse Events Leading to Permanent Discontinuation From Study Treatment and Study: Cohort 1 (Type 2 Diabetes Mellitus)
Description: \ An AE was any untoward medical occurrence in a participants or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs leading to permanent discontinuation from study were those with an AE record indicating the AE caused permanent discontinuation from the study. AEs leading to permanent discontinuation from study treatment were those AEs with an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study.
Time Frame: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 75 | 73 | 72 | 73 | 72 | 74 | 73
Participants
  Discontinuations from study due to TEAEs | 1 | 0 | 0 | 0 | 0 | 0 | 0
  Permanent discontinuations from any study intervention due to TEAEs | 0 | 3 | 11 | 10 | 5 | 17 | 5

17. Secondary Outcome: Number of Participants Reporting Adverse Events Leading to Permanent Discontinuation From Study Treatment and Study: Cohort 2 (Obesity)
Description: An AE was any untoward medical occurrence in a participants or clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. AEs leading to permanent discontinuation from study were those with an AE record indicating the AE caused permanent discontinuation from the study. AEs leading to permanent discontinuation from study treatment were those AEs with an AE record indicating that action taken with study treatment was drug withdrawn but AE did not cause the participant to be discontinued from study.
Time Frame: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 66 | 64 | 65 | 66 | 64
Participants
  Discontinuations from study due to TEAEs | 0 | 0 | 1 | 0 | 0 | 1
  Permanent discontinuations from any study intervention due to TEAEs | 5 | 12 | 19 | 15 | 24 | 22

18. Secondary Outcome: Number of Participants With Hypoglycemic Adverse Events (HAE) According to Titration Dose: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Glucose values were monitored using glucometer. Hypoglycemia =plasma/blood glucose value of <70 mg/dL (3.9 millimoles per liter [mmol/L]). Severe HAE: Participant was unable to treat him/herself due to neurological impairment (not age) and required assistance of another person, at least one neurological symptom of memory loss, confusion, uncontrolled behavior etc. Either documented blood glucose<=54 mg/dL (2.7 mmol/L). Documented symptomatic: An event during which symptoms of HAE were accompanied with plasma/blood glucose <70 mg/dL and prompt resolution with food intake, SC glucagon, or IV glucose. Probable symptomatic HAE: An event during which symptoms of an HAE were not accompanied by a plasma glucose determination but was presumably caused by a plasma glucose concentration <70 mg/dL and prompt resolution with food intake, SC glucagon, or IV glucose. Asymptomatic: An event not accompanied by typical symptoms of an HAE, but a plasma/blood glucose value of <70 mg/dL was reported.
Time Frame: Up to week 28
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Here, 'Overall Number of Participants Analyzed' signifies total number of participants with at least one dose of the given titration dose level after pooling of data across each titration dose.
Measure: Count of Participants; unit: Participants
Groups:
- Placebo (T2DM: Participants randomized to receive a single dose of PF-07081532-matching placebo QD orally.
- PF-07081532 40 mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 40 mg QD orally were included.
- PF-07081532 60mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 60 mg QD orally were included.
- PF-07081532 80 mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 80 mg QD orally were included.
- PF-07081532 120 mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 120 mg QD orally were included.
- PF-07081532 140mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 140 mg QD orally were included.
- PF-07081532 160mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 160 mg QD orally were included.
- PF-07081532 200mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 200 mg QD orally were included.
- PF-07081532 260 mg (T2DM): Participants with T2DM inadequately controlled with metformin who received PF-07081532 260 mg QD orally were included.
- Rybelsus 3mg (T2DM): Participants with T2DM inadequately controlled with metformin who received Rybelsus 3 mg QD orally were included.
- Rybelsus 7mg (T2DM): Participants with T2DM inadequately controlled with metformin who received Rybelsus 7 mg QD orally were included.
- Rybelsus 14mg (T2DM): Participants with T2DM inadequately controlled with metformin who received Rybelsus 14 mg QD orally were included.
Arm/Group | Placebo (T2DM | PF-07081532 20mg (T2DM) | PF-07081532 40 mg (T2DM) | PF-07081532 60mg (T2DM) | PF-07081532 80 mg (T2DM) | PF-07081532 120 mg (T2DM) | PF-07081532 140mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 200mg (T2DM) | PF-07081532 260 mg (T2DM) | Rybelsus 3mg (T2DM) | Rybelsus 7mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 75 | 364 | 281 | 136 | 193 | 25 | 58 | 7 | 20 | 6 | 73 | 72 | 70
Participants
  Severe Hypoglycemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Documented Symptomatic Hypoglycemia | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1
  Asymptomatic Hypoglycemia | 1 | 0 | 1 | 1 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 1 | 2
  Probable Symptomatic Hypoglycemia | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0

19. Secondary Outcome: Number of Participants With Hypoglycemic Adverse Events According to Titration Dose: Cohort 2 (Obesity)
Description: Glucose values were monitored using glucometer. Hypoglycemia =plasma/blood glucose value of <70 mg/dL (3.9 mmol/L). Severe HAE: Participant was unable to treat him/herself due to neurological impairment (not age) and required assistance of another person, at least one neurological symptom of memory loss, confusion, uncontrolled behavior etc. Either documented blood glucose<=54 mg/dL (2.7 mmol/L). Documented symptomatic: An event during which symptoms of HAE were accompanied with plasma/blood glucose <70 mg/dL u and prompt resolution with food intake, SC glucagon, or IV glucose. Probable symptomatic HAE: An event during which symptoms of an HAE were not accompanied by a plasma glucose determination but was presumably caused by a plasma glucose concentration <70 mg/dL and prompt resolution with food intake, SC glucagon, or IV glucose. Asymptomatic: An event not accompanied by typical symptoms of an HAE, but a plasma/blood glucose value of <70 mg/dL was reported.
Time Frame: Up to week 28
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Groups:
- PF-07081532 20mg (Obesity): Participants with obesity who received PF-07081532 20 mg QD orally were included.
- PF-07081532 40 mg (Obesity): Participants with obesity who received PF-07081532 40 mg QD orally were included.
- PF-07081532 60 mg (Obesity): Participants with obesity who received PF-07081532 60 mg QD orally were included.
- PF-07081532 80mg (Obesity): Participants with obesity who received PF-07081532 80 mg QD orally were included.
- PF-07081532 100 mg (Obesity): Participants with obesity who received PF-07081532 100 mg QD orally were included.
- PF-07081532 120 mg (Obesity): Participants with obesity who received PF-07081532 120 mg QD orally were included.
- PF-07081532 140mg (Obesity): Participants with obesity who received PF-07081532 140 mg QD orally were included.
- PF-07081532 160 mg (Obesity): Participants with obesity who received PF-07081532 160 mg QD orally were included.
- PF-07081532 200 mg (Obesity): Participants with obesity who received PF-07081532 200 mg QD orally were included.
- PF-07081532 260 mg (Obesity): Participants with obesity who received PF-07081532 260 mg QD orally were included.
Arm/Group | Placebo (Obesity) | PF-07081532 20mg (Obesity) | PF-07081532 40 mg (Obesity) | PF-07081532 60 mg (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 100 mg (Obesity) | PF-07081532 120 mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 160 mg (Obesity) | PF-07081532 200 mg (Obesity) | PF-07081532 260 mg (Obesity)
Number analyzed (Participants) | 64 | 325 | 310 | 170 | 220 | 56 | 43 | 140 | 47 | 121 | 28
Participants
  Severe Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Documented Symptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asymptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Probable Symptomatic Hypoglycemia | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0

20. Secondary Outcome: Number of Participants With Vital Sign Abnormalities: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Vital signs included blood pressure and pulse rate and were measured with the participants in a seated position after at least 5 minutes of rest for the participant. Criteria for abnormalities included: Systolic Blood Pressure (millimeter of mercury [mmHg]): value more than (>) 200 and value less than (<) 90; Diastolic blood pressure: value > 100 and < 40; Pulse rate: (beats per minute [BPM]): value < 40 and > 110.
Time Frame: Up to week 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Groups:
- Rybelsus 14 mg (T2DM): Participants randomized to receive Rybelsus 3 mg QD and 7 mg QD each for 4 weeks followed by 14 mg QD.
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14 mg (T2DM)
Number analyzed (Participants) | 75 | 73 | 72 | 73 | 72 | 74 | 73
Participants
  Systolic Blood Pressure (mmHg) Value <90 mmHg | 0 | 0 | 0 | 1 | 1 | 0 | 0
  Systolic Blood Pressure (mmHg) Value >200 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Value <40 mmHg | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Value >100 mmHg | 0 | 4 | 2 | 2 | 2 | 1 | 2
  Pulse Rate (bpm) Value <40 bpm | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Pulse Rate (bpm) Value >110 bpm | 0 | 1 | 1 | 0 | 0 | 1 | 0

21. Secondary Outcome: Number of Participants With Vital Sign Abnormalities: Cohort 2 (Obesity)
Description: Vital signs included blood pressure and pulse rate and were measured with the participants in a seated position after at least 5 minutes of rest for the participant. Criteria for abnormalities included: Systolic blood pressure (mmHg): value > 200 and value < 90; Diastolic blood pressure: value > 100 and < 40; Pulse rate: (BPM): value < 40 and > 110.
Time Frame: Up to week 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 66 | 64 | 65 | 66 | 64
Participants
  Systolic Blood Pressure (mmHg) Value <90 mmHg | 0 | 3 | 0 | 2 | 0 | 1
  Systolic Blood Pressure (mmHg) Value >200 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Value <40 mmHg | 0 | 0 | 0 | 0 | 0 | 0
  Diastolic Blood Pressure (mmHg) Value >100 mmHg | 4 | 4 | 4 | 0 | 2 | 3
  Pulse Rate (bpm) Value <40 bpm | 0 | 0 | 0 | 0 | 0 | 0
  Pulse Rate (bpm) Value >110 bpm | 0 | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Hematology: platelets (10^9/L)< 0.5*lower limit of normal (LLN); leukocytes< 0.6*LLN and >1.5*upper limit of normal (ULN); lymphocytes and neutrophils <0.8*LLN and >1.2*ULN; basophils, eosinophils, monocytes:>1.2*ULN; prothrombin time (sec) >1.1*ULN; prothrombin international normalized ratio >1.1*ULN; clinical chemistry: bilirubin (mg/dL), indirect bilirubin:>1.5*ULN; aspartate and alanine aminotransferase, gamma glutamyl transferase (U/L):>3.0*ULN; urea nitrogen and creatinine (mg/dL)>1.3* ULN;HDL cholesterol (mg/dL)<0.8*LLN; LDL (mg/dL)>1.2*ULN, Triglycerides (mg/dL):>1.3*ULN; Potassium (milliequivalents per liter) < 0.9*LLN and > 1.1* ULN; calcium (mg/dL)< 0.9*LLN, Thyroxine (nanograms/dL<0.8*LLN and >1.2*ULN, HbA1C (%)>1.3*ULN; Amylase, Lipase (U/L) and Glucose -Fasting (mg/dL)>1.5*ULN; urinalysis: pH> 8; urine glucose, ketones, protein, hemoglobin, nitrite and leukocyte esterase>=1. Number of participants with abnormalities in any of the laboratory parameters is reported.
Time Frame: Up to week 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 75 | 73 | 72 | 72 | 71 | 73 | 73
Participants | 67 | 64 | 57 | 57 | 61 | 59 | 64

23. Secondary Outcome: Number of Participants With Clinical Laboratory Abnormalities: Cohort 2 (Obesity)
Description: Hematology: platelets (10^9/L)< 0.5* LLN; leukocytes< 0.6*LLN and >1.5*ULN; lymphocytes and neutrophils <0.8*LLN and >1.2*ULN; basophils, eosinophils, monocytes:>1.2*ULN; prothrombin time (sec) >1.1*ULN; prothrombin international normalized ratio >1.1*ULN; clinical chemistry: bilirubin (mg/dL), indirect bilirubin:>1.5*ULN; aspartate and alanine aminotransferase, gamma glutamyl transferase (U/L):>3.0*ULN; urea nitrogen and creatinine (mg/dL)>1.3* ULN;HDL cholesterol (mg/dL)<0.8*LLN; LDL (mg/dL)>1.2*ULN, Triglycerides (mg/dL):>1.3*ULN; Potassium (milliequivalents per liter) < 0.9*LLN and > 1.1* ULN; calcium (mg/dL)< 0.9*LLN, Thyroxine (nanograms/dL<0.8*LLN and >1.2*ULN, HbA1C (%)>1.3*ULN; Amylase, Lipase (U/L) and Glucose -Fasting (mg/dL)>1.5*ULN; urinalysis: pH> 8; urine glucose, ketones, protein, hemoglobin, nitrite and leukocyte esterase>=1. Number of participants with abnormalities in any of the laboratory parameters is reported.
Time Frame: Up to week 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 63 | 63 | 63 | 66 | 64
Participants | 36 | 31 | 40 | 40 | 48 | 36

24. Secondary Outcome: Number of Participants With ECG Abnormalities: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Standard 12-lead ECGs were performed after the participant had rested quietly for more than 10 minutes in a supine position utilizing an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, QT interval corrected using Fridericia's formula (QTcF), and QRS complex. ECG abnormalities were categorized as: PR interval (milliseconds [msec]), Value >= 300; percent change (%Chg) greater than equal (>=) 25/50%. QRS duration (msec): Value >= 140 and %Chg >= 50%. QT interval (msec): Value > 500; QTCF interval (msec): 450 < Value <= 480, 480 < Value <= 500, Value > 500; 30 <= Change (Chg) <= 60; Chg > 60.
Time Frame: Up to week 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 75 | 73 | 72 | 73 | 72 | 74 | 73
Participants
  PR Interval, (MSEC) value >=300 | 1 | 0 | 0 | 1 | 0 | 0 | 0
  PR Interval, (MSEC) %Chg >= 25/50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QRS duration, (MSEC) value >=140 | 1 | 0 | 0 | 1 | 0 | 0 | 3
  QRS duration, (MSEC) %Chg >=50% | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QT interval, single beat (MSEC) value > 500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF interval, single beat (MSEC) 450 < Value <=480 | 5 | 7 | 3 | 5 | 5 | 2 | 5
  QTCF interval, single beat (MSEC) 480 < Value <=500 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  QTCF interval, single beat (MSEC) Value > 500 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF interval, single beat (MSEC) 30 <= Chg <= 60 | 3 | 7 | 5 | 4 | 3 | 10 | 8
  QTCF interval, single beat (MSEC) Chg > 60 | 0 | 0 | 0 | 0 | 0 | 0 | 0

25. Secondary Outcome: Number of Participants With ECG Abnormalities: Cohort 2 (Obesity)
Description: Standard 12-lead ECGs were performed after the participant had rested quietly for more than 10 minutes in a supine position utilizing an ECG machine that automatically calculated the heart rate and measured PR interval, QT interval, QTcF, and QRS complex. ECG abnormalities were categorized as: PR interval msec, Value >= 300; percentage change (%Chg) >= 25/50%. QRS duration (msec): Value >= 140 and %Chg >= 50%. QT interval (msec): Value > 500; QTCF interval (msec): 450 < Value <= 480, 480 < Value <= 500, Value > 500; 30 <= Change (Chg) <= 60; Chg > 60.
Time Frame: Up to week 28
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 66 | 64 | 65 | 66 | 64
Participants
  PR Interval, (MSEC) value >=300 | 0 | 0 | 0 | 0 | 1 | 0
  PR Interval, (MSEC) %Chg >= 25/50% | 0 | 0 | 0 | 0 | 1 | 0
  QRS duration, (MSEC) value >=140 | 1 | 0 | 0 | 0 | 0 | 0
  QRS duration, (MSEC) %Chg >=50% | 0 | 0 | 0 | 0 | 0 | 0
  QT interval, single beat (MSEC) value > 500 | 0 | 0 | 0 | 1 | 0 | 0
  QTCF interval, single beat (MSEC) 450 < Value <=480 | 9 | 3 | 4 | 2 | 4 | 7
  QTCF interval, single beat (MSEC) 480 < Value <=500 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF interval, single beat (MSEC) Value > 500 | 0 | 0 | 0 | 0 | 0 | 0
  QTCF interval, single beat (MSEC) 30 <= Chg <= 60 | 3 | 8 | 4 | 4 | 4 | 3
  QTCF interval, single beat (MSEC) Chg > 60 | 0 | 0 | 0 | 0 | 0 | 0

26. Secondary Outcome: Number of Participants According to Columbia-Suicide Severity Rating Scale (C-SSRS) Category: Cohort 2 (Obesity) Only
Description: C-SSRS is an interview-based rating scale to assess suicidal ideation and suicidal behavior and had a binary response (yes/no). C-SSRS data was mapped to C-CASA per Guidance for Industry: Suicidal Ideation and Behavior: Prospective Assessment of Occurrence in Clinical Trials. A participant was said to have suicidal behavior in case of any of following events: 1) completed suicide; 2) suicide attempt; or 3) preparatory acts toward imminent suicidal behavior. A participant showed suicidal ideation if they responded 'yes' to any of the 5 questions, 'Wish to be dead; Non-Specific Active Suicidal Thoughts Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent. The participant was said to exhibit Self-injurious behavior, no suicidal intent if they responded as Yes to 'Has participant engaged in Non-suicidal Self-Injurious Behavior
Time Frame: Baseline (result closest prior to dosing on Day 1), anytime post-baseline (Up to Week 28)
Population: Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to the product they actually received. This outcome measure was planned to be assessed in Cohort 2 only.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 64 | 66 | 64 | 65 | 66 | 64
Participants
  Baseline: <1> Completed suicide | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: <2> Suicide attempt | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: <3> Preparatory acts towards imminent suicidal behavior | 0 | 0 | 0 | 0 | 0 | 0
  Baseline: <4> Suicidal ideation | 0 | 0 | 0 | 0 | 0 | 1
  Baseline: <7> Self-injurious behavior, no suicidal intent | 0 | 0 | 0 | 0 | 0 | 0
  Post-Baseline: <1> Completed suicide | 0 | 0 | 0 | 0 | 0 | 0
  Post-Baseline: <2> Suicide attempt | 0 | 0 | 0 | 0 | 0 | 0
  Post-Baseline: <3> Preparatory acts towards imminent suicidal behavior | 1 | 0 | 0 | 0 | 0 | 0
  Post-Baseline: <4> Suicidal ideation | 0 | 0 | 0 | 0 | 0 | 1
  Post-Baseline: <7> Self-injurious behavior, no suicidal intent | 1 | 0 | 0 | 0 | 0 | 0

27. Other Pre Specified Outcome: Placebo-adjusted, Change From Baseline in Percentage of Glycated Hemoglobin (HbA1c) at Week 16: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Analysis was performed using mixed model repeated measures (MMRM) model including treatment, gender strata and time as fixed effects, baseline*time interaction, time*treatment interaction, and baseline as a covariate with time fitted as a repeated effect and participant as a random effect.
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 16
Population: Evaluable set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to randomized intervention. Here, "Overall Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1c
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 24 | 30 | 21 | 22 | 25 | 21 | 24
Percentage of HbA1c | -0.07 (0.109) | -1.03 (0.106) | -1.37 (0.112) | -1.44 (0.111) | -1.34 (0.110) | -1.36 (0.114) | -0.94 (0.109)
Statistical Analysis 1: Comparison: Placebo (T2DM) vs PF-07081532 20mg (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -0.95, 90% CI 2-sided [-1.20 to -0.70]
Statistical Analysis 2: Comparison: Placebo (T2DM) vs PF-07081532 40mg (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.30, 90% CI 2-sided [-1.55 to -1.04]
Statistical Analysis 3: Comparison: Placebo (T2DM) vs PF-07081532 80mg (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.37, 90% CI [-1.62 to -1.11]
Statistical Analysis 4: Comparison: Placebo (T2DM) vs PF-07081532 160mg (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.26, 90% CI 2-sided [-1.52 to -1.01]
Statistical Analysis 5: Comparison: Placebo (T2DM) vs PF-07081532 260mg (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -1.29, 90% CI [-1.55 to -1.03]
Statistical Analysis 6: Comparison: Placebo (T2DM) vs Rybelsus 14mg (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -0.86, 90% CI 2-sided [-1.12 to -0.61]

28. Other Pre Specified Outcome: Placebo-adjusted, Percent Change From Baseline in Body Weight at Week 20: Cohort 2 (Obesity)
Description: Body weight was measured using a calibrated weighing scale. Analysis was performed using MMRM model including treatment, gender strata and time as fixed effects, baseline*time interaction, time*treatment interaction, and baseline as a covariate with time fitted as a repeated effect and participant as a random effect.
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 20
Population: as for outcome 27
Measure: Least Squares Mean (Standard Error); unit: Percent change
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 45 | 44 | 37 | 38 | 31 | 28
Percent change | -1.84 (0.612) | -4.28 (0.623) | -6.21 (0.654) | -7.47 (0.628) | -6.88 (0.638) | -7.26 (0.664)
Statistical Analysis 1: Comparison: Placebo (Obesity) vs PF-07081532 80mg (Obesity); Test type: Other; p = 0.0055, Mixed Models Analysis; LS Mean Difference = -2.44, 90% CI 2-sided [-3.88 to -1.00]
Statistical Analysis 2: Comparison: Placebo (Obesity) vs PF-07081532 140mg (Obesity); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -4.37, 90% CI 2-sided [-5.84 to -2.89]
Statistical Analysis 3: Comparison: Placebo (Obesity) vs PF-07081532 200mg (Obesity,5 Steps); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -5.63, 90% CI 2-sided [-7.07 to -4.18]
Statistical Analysis 4: Comparison: Placebo (Obesity) vs PF-07081532 200mg (Obesity,4 Steps); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -5.04, 90% CI 2-sided [-6.50 to -3.58]
Statistical Analysis 5: Comparison: Placebo (Obesity) vs PF-07081532 260mg (Obesity); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -5.42, 90% CI 2-sided [-6.91 to -3.93]

29. Other Pre Specified Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 16: Cohort 1 (Type 2 Diabetes Mellitus)
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 16
Population: Evaluable set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to randomized intervention. Here, "Number of Participants Analyzed" refers to participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Milligrams per deciliter
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 24 | 30 | 21 | 22 | 25 | 21 | 24
Milligrams per deciliter | 160.70 (39.595) | 135.59 (31.746) | 127.00 (35.928) | 132.19 (31.541) | 127.65 (28.839) | 125.07 (46.924) | 130.06 (28.120)

30. Other Pre Specified Outcome: Percent Change From Baseline in Body Weight at Week 16: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Body weight was measured using a calibrated weighing scale.
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 16
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM)
Number analyzed (Participants) | 29 | 32 | 30 | 28 | 28 | 30 | 27
Percent change | 93.164 (22.0659) | 86.251 (17.3464) | 91.556 (23.4071) | 92.979 (24.5045) | 85.564 (17.9582) | 87.658 (21.6950) | 91.799 (20.4605)

31. Other Pre Specified Outcome: Placebo-adjusted, Change From Baseline in Percentage of HbA1C in the Rybelsus Arm Versus Placebo Arm at Week 16: Cohort 1 (Type 2 Diabetes Mellitus)
Description: Analysis was performed using MMRM model including treatment, gender strata and time as fixed effects, baseline*time interaction, time*treatment interaction, and baseline as a covariate with time fitted as a repeated effect and participant as a random effect. This outcome measure was planned to be analyzed only for rybelsus arm and placebo arm as pre-specified in the protocol.
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 16
Population: Evaluable set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to randomized intervention.
Measure: Least Squares Mean (Standard Error); unit: Percentage of HbA1C
Arm/Group | Rybelsus 14mg (T2DM) | Placebo (T2DM)
Number analyzed (Participants) | 24 | 24
Percentage of HbA1C | -0.94 (0.109) | -0.07 (0.109)
Statistical Analysis 1: Comparison: Rybelsus 14mg (T2DM) vs Placebo (T2DM); Test type: Other; p < .0001, Mixed Models Analysis; LS Mean Difference = -0.86, 90% CI 2-sided [-1.12 to -0.61]

32. Other Pre Specified Outcome: Absolute Change From Baseline in Waist Circumference at Week 12 and 24: Cohort 2 (Obesity)
Description: Waist circumference was measured at midpoint, between lower margin of last palpable rib and top of iliac crest (approximately 1 inch [2.54 cm] above the navel). It was measured by using an anthropometric tape (stretch-resistant).
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], Week 12, 24
Population: Evaluable set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention. Participants were analyzed according to randomized intervention. Here "Number Analyzed" refers to the number of participants evaluable for the specified rows.
Measure: Mean (Standard Deviation); unit: Centimeter
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 57 | 53 | 49 | 56 | 53 | 50
Centimeter
  Week 12 | -2.702 (4.1726) | -2.574 (5.0872) | -3.017 (5.9117) | -3.559 (6.5122) | -2.191 (5.2942) | -1.079 (4.6710)
  Week 24: number analyzed (Participants) | 12 | 12 | 11 | 9 | 7 | 4
  Week 24 | -4.233 (5.3953) | -5.147 (4.1807) | -6.314 (10.2170) | -2.722 (7.6706) | -10.297 (7.7652) | -6.450 (4.2123)

33. Other Pre Specified Outcome: Absolute Change From Baseline in Waist-to-hip Ratio at Week 12 and Week 24: Cohort 2 (Obesity)
Description: as for outcome 9
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], week 12, 24
Population: as for outcome 32
Measure: Mean (Standard Deviation); unit: Ratio
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 57 | 53 | 49 | 56 | 53 | 50
Ratio
  Week 12 | -0.013 (0.0374) | -0.002 (0.0459) | -0.006 (0.0578) | -0.010 (0.0683) | -0.002 (0.0423) | 0.015 (0.0557)
  Week 24: number analyzed (Participants) | 12 | 12 | 11 | 9 | 7 | 4
  Week 24 | -0.023 (0.0419) | -0.017 (0.0250) | -0.032 (0.0588) | 0.018 (0.0563) | -0.009 (0.0498) | -0.037 (0.0574)

34. Other Pre Specified Outcome: Change From Baseline in Homeostatic Model Assessment for Insulin Resistance (HOMA-IR) at Week 16: Cohort 2 (Obesity)
Description: HOMA-IR was calculated as: ([FPI]*(FPG)/405 in terms of Mg/dL* (milliunits per liter).
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 16
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Milliunits per liter
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 53 | 48 | 42 | 46 | 42 | 39
Milliunits per liter | 0.630 (2.1753) | 0.185 (2.0579) | -0.121 (4.7540) | 0.984 (3.9090) | -1.172 (2.7360) | -0.210 (1.1373)

35. Other Pre Specified Outcome: Change From Baseline in Homeostatic Model Assessment for Insulin Sensitivity (HOMA-S) at Week 16: Cohort 2 (Obesity)
Description: HOMA-S was calculated as (22.5/[FPI]*FPG)) *100 and measured in terms of. percentage sensitivity.
Time Frame: Baseline [(Baseline is defined as the result closest prior to dosing at Visit 3 (Day 1)], at Week 16
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Percentage sensitivity
Arm/Group | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
Number analyzed (Participants) | 53 | 48 | 42 | 46 | 42 | 39
Percentage sensitivity | -2.419 (51.8526) | 1.594 (24.1848) | 7.807 (26.5041) | -7.085 (21.6406) | 3.497 (68.2570) | -2.045 (28.8973)

ADVERSE EVENTS:
Time Frame: Part1 and 2: From start of treatment up to minimum of 28 days after last dose of treatment administration (maximum up to Week 28)
Description: Same event may appear as both non-SAE and SAE. What is presented are distinct events. An event may be categorized as serious in 1 participant and non-serious in other participant, or a participant may have experienced both SAE and non-SAE. Safety analysis set included all participants randomly assigned to study intervention and who took at least 1 dose of study intervention.
Arm/Group | Placebo (T2DM) | PF-07081532 20mg (T2DM) | PF-07081532 40mg (T2DM) | PF-07081532 80mg (T2DM) | PF-07081532 160mg (T2DM) | PF-07081532 260mg (T2DM) | Rybelsus 14mg (T2DM) | Placebo (Obesity) | PF-07081532 80mg (Obesity) | PF-07081532 140mg (Obesity) | PF-07081532 200mg (Obesity,5 Steps) | PF-07081532 200mg (Obesity,4 Steps) | PF-07081532 260mg (Obesity)
All-Cause Mortality (participants affected / at risk) | 1/75 | 0/73 | 0/72 | 0/73 | 0/72 | 0/74 | 0/73 | 0/64 | 0/66 | 0/64 | 0/65 | 0/66 | 0/64
Serious Adverse Events (participants affected / at risk) | 1/75 | 0/73 | 3/72 | 3/73 | 1/72 | 2/74 | 1/73 | 1/64 | 2/66 | 2/64 | 1/65 | 2/66 | 2/64
Other Adverse Events (participants affected / at risk) | 23/75 | 31/73 | 46/72 | 37/73 | 41/72 | 51/74 | 32/73 | 42/64 | 50/66 | 48/64 | 55/65 | 59/66 | 53/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (T2DM) (N=75) | PF-07081532 20mg (T2DM) (N=73) | PF-07081532 40mg (T2DM) (N=72) | PF-07081532 80mg (T2DM) (N=73) | PF-07081532 160mg (T2DM) (N=72) | PF-07081532 260mg (T2DM) (N=74) | Rybelsus 14mg (T2DM) (N=73) | Placebo (Obesity) (N=64) | PF-07081532 80mg (Obesity) (N=66) | PF-07081532 140mg (Obesity) (N=64) | PF-07081532 200mg (Obesity,5 Steps) (N=65) | PF-07081532 200mg (Obesity,4 Steps) (N=66) | PF-07081532 260mg (Obesity) (N=64)
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sepsis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gout (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Cardiac arrest (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test abnormal (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Carcinoid tumour (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Allergic respiratory symptom (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (T2DM) (N=75) | PF-07081532 20mg (T2DM) (N=73) | PF-07081532 40mg (T2DM) (N=72) | PF-07081532 80mg (T2DM) (N=73) | PF-07081532 160mg (T2DM) (N=72) | PF-07081532 260mg (T2DM) (N=74) | Rybelsus 14mg (T2DM) (N=73) | Placebo (Obesity) (N=64) | PF-07081532 80mg (Obesity) (N=66) | PF-07081532 140mg (Obesity) (N=64) | PF-07081532 200mg (Obesity,5 Steps) (N=65) | PF-07081532 200mg (Obesity,4 Steps) (N=66) | PF-07081532 260mg (Obesity) (N=64)
Abdominal distension (Gastrointestinal disorders) | 0 | 1 | 5 | 2 | 2 | 1 | 1 | 4 | 2 | 3 | 1 | 3 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 5 | 1 | 1 | 2 | 2 | 4 | 3 | 6 | 2 | 10 | 4
Abdominal pain upper (Gastrointestinal disorders) | 0 | 3 | 5 | 1 | 1 | 1 | 1 | 1 | 1 | 4 | 6 | 3 | 3
Constipation (Gastrointestinal disorders) | 1 | 2 | 7 | 3 | 4 | 6 | 4 | 5 | 14 | 15 | 15 | 23 | 17
Diarrhoea (Gastrointestinal disorders) | 1 | 8 | 9 | 8 | 4 | 8 | 6 | 12 | 10 | 10 | 16 | 17 | 17
Dyspepsia (Gastrointestinal disorders) | 1 | 3 | 2 | 4 | 4 | 3 | 2 | 2 | 6 | 4 | 6 | 9 | 4
Eructation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 2 | 4 | 5
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 2 | 3 | 4 | 3 | 1 | 1 | 10 | 6 | 5 | 13 | 6
Nausea (Gastrointestinal disorders) | 3 | 11 | 17 | 21 | 14 | 19 | 10 | 8 | 34 | 30 | 38 | 40 | 32
Vomiting (Gastrointestinal disorders) | 1 | 1 | 6 | 11 | 6 | 11 | 6 | 1 | 7 | 10 | 21 | 19 | 22
Fatigue (General disorders) | 0 | 0 | 4 | 1 | 2 | 2 | 2 | 5 | 7 | 5 | 6 | 5 | 5
COVID-19 (Infections and infestations) | 0 | 2 | 0 | 1 | 1 | 2 | 0 | 5 | 3 | 2 | 1 | 2 | 5
Nasopharyngitis (Infections and infestations) | 1 | 0 | 3 | 2 | 1 | 2 | 0 | 0 | 5 | 2 | 4 | 2 | 4
Urinary tract infection (Infections and infestations) | 1 | 1 | 4 | 1 | 0 | 6 | 4 | 2 | 2 | 2 | 6 | 5 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 1 | 5 | 3 | 4 | 7 | 0 | 5 | 5 | 7 | 3 | 8 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 1 | 1 | 0 | 1 | 1 | 2 | 2 | 1 | 3 | 4 | 3
Dizziness (Nervous system disorders) | 2 | 0 | 1 | 1 | 2 | 7 | 0 | 3 | 4 | 2 | 1 | 4 | 4
Headache (Nervous system disorders) | 0 | 2 | 5 | 2 | 1 | 1 | 2 | 5 | 7 | 4 | 7 | 9 | 5
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2 | 0 | 1 | 2 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 5 | 6 | 1 | 0 | 3 | 1 | 3 | 2 | 3
Flatulence (Gastrointestinal disorders) | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 2 | 1 | 1 | 1 | 3 | 4
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 3 | 1 | 2 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 1 | 4 | 1 | 3 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 0 | 3 | 1 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 1 | 0 | 1 | 0 | 3 | 3 | 2 | 1 | 4 | 5 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 2 | 0 | 2 | 1 | 2 | 1 | 4 | 1
Lipase increased (Investigations) | 0 | 3 | 4 | 1 | 0 | 3 | 3 | 0 | 2 | 0 | 0 | 1 | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 6 | 1 | 1 | 1 | 1 | 1 | 3 | 0 | 0 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 1
Gastrititis (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Chest discomfort (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 1
Early satiety (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 2
Pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Ear infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 2 | 1 | 1 | 3 | 2 | 1
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Pharyngitis (Infections and infestations) | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Viral infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Amylase increased (Investigations) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 3 | 1
Hepatic enzyme increased (Investigations) | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 1 | 2 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 1 | 1 | 1 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 3 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Head discomfort (Nervous system disorders) | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Migraine (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Microalbuminuria (Renal and urinary disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 1 | 1 | 1
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 2 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 2 | 1 | 1 | 2 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Hypotension (Vascular disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 1
Ventricular extrasystoles (Cardiac disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 2 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
1 participant in placebo (T2DM) arm with withdrawal reason as Death in treatment phase was also counted in follow-up with the reason for discontinuation as death since exact date of last dose was unknown.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2022-09-13): https://cdn.clinicaltrials.gov/large-docs/77/NCT05579977/Prot_000.pdf
  • Statistical Analysis Plan (2023-09-27): https://cdn.clinicaltrials.gov/large-docs/77/NCT05579977/SAP_001.pdf